CLINICAL TRIAL: NCT01928862
Title: A Randomized, Assessor-Blind, Multicenter, Dose-Ranging Study Comparing the Safety and Efficacy of Prepopik® Versus Polyethylene Glycol Preparation (Local Standard of Care) in Children Aged 9 Years to 16 Years
Brief Title: Efficacy and Safety of Prepopik® in Children for Overall Colon Cleansing in Preparation for Colonoscopy
Acronym: Prepopik PREA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000103
Record Dates: First submitted 2013-08-19; First posted 2013-08-27 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-03

CONDITIONS: Need for Bowel Preparation
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Prepopik® ½ Sachet x 2 (9-12 years) (Experimental): Prepopik® ½ Sachet x 2 (9-12 years)
  Interventions: Drug: Prepopik® ½ Sachet x 2 (9-12 years)
- Prepopik® 1 Sachet x 2 (9-12 years) (Experimental): Prepopik® 1 Sachet x 2 (9-12 years)
  Interventions: Drug: Prepopik® 1 Sachet x 2 (9-12 years)
- Oral polyethylene glycol (PEG) based preparation (9-12 years) (Active Comparator): Local standard of care
  Interventions: Drug: Oral polyethylene glycol (PEG) based preparation (9-12 years)
- Prepopik® 1 Sachet x 2 (13-16 years) (Experimental): Prepopik® 1 Sachet x 2 (13-16 years)
  Interventions: Drug: Prepopik® 1 Sachet x 2 (13-16 years)
- Oral polyethylene glycol (PEG) based preparation (13-16 years) (Active Comparator): Local standard of care
  Interventions: Drug: Oral polyethylene glycol (PEG) based preparation (13-16 years)

INTERVENTIONS:
Drug: Prepopik® ½ Sachet x 2 (9-12 years)
  Other Names: Prepopik®
  Arms: Prepopik® ½ Sachet x 2 (9-12 years)
Drug: Prepopik® 1 Sachet x 2 (9-12 years)
  Other Names: Prepopik®
  Arms: Prepopik® 1 Sachet x 2 (9-12 years)
Drug: Oral polyethylene glycol (PEG) based preparation (9-12 years)
  Arms: Oral polyethylene glycol (PEG) based preparation (9-12 years)
Drug: Prepopik® 1 Sachet x 2 (13-16 years)
  Other Names: Prepopik®
  Arms: Prepopik® 1 Sachet x 2 (13-16 years)
Drug: Oral polyethylene glycol (PEG) based preparation (13-16 years)
  Arms: Oral polyethylene glycol (PEG) based preparation (13-16 years)

SUMMARY:
To study the efficacy and safety of Prepopik® in children aged 9 to 16 years for overall colon cleansing in preparation of colonoscopy

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 9 years to 16 years, inclusive, being scheduled to undergo elective colonoscopy
* Subjects must have had 3 or more spontaneous bowel movements per week for 1 month prior to the colonoscopy
* Female subjects of childbearing potential must undergo a pregnancy test at screening and again at randomization

Exclusion Criteria:

* Acute surgical abdominal conditions (e.g., acute obstruction or perforation)
* Hospitalized for inflammatory bowel disease
* Any prior colorectal surgery, excluding appendectomy, hemorrhoid surgery, or prior endoscopic surgical procedures
* Colon disease (history of colonic cancer, toxic megacolon, toxic colitis, idiopathic pseudo obstruction, hypomotility syndrome, colon resection)
* Ascites
* Gastrointestinal disorder (active ulcer, outlet obstruction, retention, gastroparesis, ileus)
* Upper gastrointestinal surgery (gastric resection, gastric banding, gastric bypass)
* Significant cardiovascular disease as determined by the investigator
* If subject has a history of renal insufficiency, serum creatinine and potassium must be within normal limits
* Any clinically significant laboratory value at screening, including pre- existing electrolyte abnormality, based on clinical history
* Hypersensitivity to active ingredients

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2014-06-03 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (9):
- United States (9):
  - University of Alabama, Birmingham, Alabama
  - University California San Diego - Rady's Children's Hospital, San Diego, California
  - IU Medical Center / Riley Hospital, Indianapolis, Indiana
  - John Hopkins, Baltimore, Maryland
  - Stony Brook Children's, Stony Brook, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 9 investigative sites in the United States (US).
Pre-assignment Details: Eighty participants were screened out of which 78 participants were randomized in this trial. Two were screening failures (participant not fulfilling inclusion/exclusion criteria [n=1], other [n=1]).
Groups:
- Prepopik® ½ Sachet x 2 (9-12 Years): Prepopik® (sodium picosulfate 10 mg; magnesium oxide 3.5 g and anhydrous citric acid 12 g) reconstituted with water was administered in "Split Dose" method. The first dose was administered between 5:00 PM and 9:00 PM on the day before the colonoscopy procedure. The second dose was given on the next day, at least 6 hours after the first dose and approximately 5 hours before but no more than 9 hours prior to the colonoscopy.
  "Day Before" method was the alternative method if "Split Dose" was not appropriate. In "Day Before" method, the first dose was administered during the afternoon or early evening before the colonoscopy and the second dose was administered 6 hours later during the evening before the colonoscopy.
  The dose was ½ sachet for this subset of participants (9-12 years old).
- Prepopik® 1 Sachet x 2 (9-12 Years): Prepopik® (sodium picosulfate 10 mg; magnesium oxide 3.5 g and anhydrous citric acid 12 g) reconstituted with water was administered in "Split Dose" method. The first dose was administered between 5:00 PM and 9:00 PM on the day before the colonoscopy procedure. The second dose was given on the next day, at least 6 hours after the first dose and approximately 5 hours before but no more than 9 hours prior to the colonoscopy.
  "Day Before" method was the alternative method if "Split Dose" was not appropriate. In "Day Before" method, the first dose was administered during the afternoon or early evening before the colonoscopy and the second dose was administered 6 hours later during the evening before the colonoscopy.
  The dose was 1 sachet for this subset of participants (9-12 years old).
- Oral Polyethylene Glycol (PEG) Based Preparation (9-12 Years): Oral PEG based preparation/ local standard of care following appropriate label and/or institutional instructions for this subset of participants (9-12 years old).
- Prepopik® 1 Sachet x 2 (13-16 Years): Prepopik® (sodium picosulfate 10 mg; magnesium oxide 3.5 g and anhydrous citric acid 12 g) reconstituted with water was administered in "Split Dose" method. The first dose was administered between 5:00 PM and 9:00 PM on the day before the colonoscopy procedure. The second dose was given on the next day, at least 6 hours after the first dose and approximately 5 hours before but no more than 9 hours prior to the colonoscopy.
  "Day Before" method was the alternative method if "Split Dose" was not appropriate. In "Day Before" method, the first dose was administered during the afternoon or early evening before the colonoscopy and the second dose was administered 6 hours later during the evening before the colonoscopy.
  The dose was 1 sachet for this subset of participants (13-16 years old).
- Oral Polyethylene Glycol (PEG) Based Preparation (13-16 Years): Oral PEG based preparation/ local standard of care following appropriate label and/or institutional instructions for this subset of participants (13-16 years old).
Period: Overall Study
Arm/Group | Prepopik® ½ Sachet x 2 (9-12 Years) | Prepopik® 1 Sachet x 2 (9-12 Years) | Oral Polyethylene Glycol (PEG) Based Preparation (9-12 Years) | Prepopik® 1 Sachet x 2 (13-16 Years) | Oral Polyethylene Glycol (PEG) Based Preparation (13-16 Years)
Started | 16 | 16 | 16 | 16 | 14
Completed | 15 | 16 | 16 | 16 | 13
Not Completed | 1 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prepopik® ½ Sachet x 2 (9-12 Years) | Prepopik® 1 Sachet x 2 (9-12 Years) | Oral Polyethylene Glycol (PEG) Based Preparation (9-12 Years) | Prepopik® 1 Sachet x 2 (13-16 Years) | Oral Polyethylene Glycol (PEG) Based Preparation (13-16 Years) | Total
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 14 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.8 (1.00) | 10.5 (1.21) | 10.4 (1.20) | 15.0 (1.03) | 14.9 (0.92) | 12.2 (2.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 8 | 11 | 11 | 53
  Male | 5 | 4 | 8 | 5 | 3 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 1 | 0 | 4
  Not Hispanic or Latino | 16 | 14 | 15 | 15 | 14 | 74
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 5 | 1 | 0 | 6
  White | 15 | 16 | 11 | 15 | 14 | 71
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Defined by "Excellent" or "Good" in the Aronchick Scale
Description: Aronchick scale is a 4-point scale that grades colon cleansing as Excellent (>90% of mucosa seen, mostly liquid stool, minimal suctioning needed for adequate visualization), Good (>90% of mucosa seen, mostly liquid stool, significant suctioning needed for adequate visualization), Fair (>90% of mucosa seen, mixture of liquid and semisolid stool, could be suctioned and/or washed) or Inadequate (<90% of mucosa seen, mixture of semisolid and solid stool which could not be suctioned or washed). The participant is considered to be a responder if overall colon cleansing is "excellent" or "good" on this 4-point scale.
Time Frame: On the day of colonoscopy
Population: The primary efficacy analysis was based on the intention-to-treat (ITT) analysis set, which included all participants who were randomized.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Prepopik® ½ Sachet x 2 (9-12 Years) | Prepopik® 1 Sachet x 2 (9-12 Years) | Oral Polyethylene Glycol (PEG) Based Preparation (9-12 Years) | Prepopik® 1 Sachet x 2 (13-16 Years) | Oral Polyethylene Glycol (PEG) Based Preparation (13-16 Years)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 14
percentage of participants | 50 [27.9 to 72.1] | 87.5 [65.6 to 97.7] | 81.3 [58.3 to 94.7] | 81.3 [58.3 to 94.7] | 85.7 [61.5 to 97.4]
Statistical Analysis 1: Comparison: Prepopik® ½ Sachet x 2 (9-12 Years) vs Oral Polyethylene Glycol (PEG) Based Preparation (9-12 Years); Confidence interval (CI) of the difference in proportions between each Prepopik® group and PEG within each age group was calculated using the Clopper-Pearson method; Test type: Other; Treatment difference = -31.3, 90% CI 2-sided [-58.8 to 0.8]
Statistical Analysis 2: Comparison: Prepopik® 1 Sachet x 2 (9-12 Years) vs Oral Polyethylene Glycol (PEG) Based Preparation (9-12 Years); CI of the difference in proportions between each Prepopik® group and PEG within each age group was calculated using the Clopper-Pearson method; Test type: Other; Treatment Difference = 6.3, 90% CI 2-sided [-25.3 to 36.9]
Statistical Analysis 3: Comparison: Prepopik® 1 Sachet x 2 (13-16 Years) vs Oral Polyethylene Glycol (PEG) Based Preparation (13-16 Years); [analysis description as in outcome 1, analysis 2]; Test type: Other; Treatment Difference = -4.5, 90% CI 2-sided [-33.5 to 26.3]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant taking part in a clinical trial. Proportion of participants with AE are presented.
Time Frame: Up to 33 days after colonoscopy
Population: The safety analysis set included participants who received at least one dose of the trial medication. Participants were analyzed according to actual treatment received. One of the participant randomized to Prepopik® ½ sachet x 2 (9-12 years) received Prepopik® 1 sachet x 2 (9-12 years) instead (n=17).
Measure: Number; unit: participants
Arm/Group | Prepopik® ½ Sachet x 2 (9-12 Years) | Prepopik® 1 Sachet x 2 (9-12 Years) | Oral Polyethylene Glycol (PEG) Based Preparation (9-12 Years) | Prepopik® 1 Sachet x 2 (13-16 Years) | Oral Polyethylene Glycol (PEG) Based Preparation (13-16 Years)
Number analyzed (Participants) | 15 | 17 | 15 | 16 | 12
participants | 8 | 5 | 6 | 10 | 11

3. Secondary Outcome: Number of Participants With Abnormal Findings in Laboratory Tests
Description: Proportion of participants with abnormal findings in laboratory tests are presented.
Time Frame: From up to 42 days prior to colonoscopy, at the day of colonoscopy, and up to 7 days post colonoscopy
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Prepopik® ½ Sachet x 2 (9-12 Years) | Prepopik® 1 Sachet x 2 (9-12 Years) | Oral Polyethylene Glycol (PEG) Based Preparation (9-12 Years) | Prepopik® 1 Sachet x 2 (13-16 Years) | Oral Polyethylene Glycol (PEG) Based Preparation (13-16 Years)
Number analyzed (Participants) | 15 | 17 | 15 | 16 | 12
participants
  Basophils (ratio) ≥upper limit (≥1) | 2 | 2 | 4 | 1 | 1
  Eosinophils (ratio) ≥upper limit (≥5) | 4 | 1 | 3 | 2 | 1
  Erythrocytes (×10^12/L)≤ lower limit(≤3.5×10^12/L) | 0 | 1 | 0 | 0 | 0
  Leukocytes (×10^9/L) ≤lower limit (≤4×10^9/L) | 1 | 2 | 1 | 1 | 2
  Lymphocytes (×10^9/L) ≤lower limit (≤1×10^9/L) | 0 | 0 | 1 | 1 | 1
  Monocytes (ratio) ≥upper limit (≥5) | 0 | 0 | 0 | 1 | 0
  Neutrophils (×10^9/L) ≥upper limit (≥10×10^9/L) | 0 | 0 | 0 | 0 | 1
  Bilirubin (μmol/L) ≥upper limit (≥34 μmol/L) | 1 | 0 | 0 | 0 | 0
  Glucose (mmol/L) ≤lower limit (≤2.8 mmol/L) | 0 | 1 | 0 | 1 | 1
  Protein (g/L) ≥upper limit (≥80 g/L) | 2 | 1 | 0 | 2 | 2

4. Secondary Outcome: Number of Participants With Abnormal Findings in Physical Examination
Description: Complete physical examination was conducted at screening and directed physical examinations at other time-points. Directed physical examinations are presented.
Time Frame: From up to 42 days prior to colonoscopy, on the day of randomization, and at the day of colonoscopy
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- Oral Polyethylene Glycol (PEG) Based Preparation (9-12 Years): Oral PEG preparation/ local standard of care following appropriate label and/or institutional instructions for this subset of participants (9-12 years old).
Arm/Group | Prepopik® ½ Sachet x 2 (9-12 Years) | Prepopik® 1 Sachet x 2 (9-12 Years) | Oral Polyethylene Glycol (PEG) Based Preparation (9-12 Years) | Prepopik® 1 Sachet x 2 (13-16 Years) | Oral Polyethylene Glycol (PEG) Based Preparation (13-16 Years)
Number analyzed (Participants) | 15 | 17 | 15 | 16 | 12
participants | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants Who Took the Assigned Dose for Colon Cleansing
Description: The proportion of participants who took the assigned dose of Prepopik® was assessed.
Time Frame: Approx. 1 day (From the day before colonoscopy to the day of colonoscopy)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Prepopik® ½ Sachet x 2 (9-12 Years) | Prepopik® 1 Sachet x 2 (9-12 Years) | Oral Polyethylene Glycol (PEG) Based Preparation (9-12 Years) | Prepopik® 1 Sachet x 2 (13-16 Years) | Oral Polyethylene Glycol (PEG) Based Preparation (13-16 Years)
Number analyzed (Participants) | 15 | 17 | 15 | 16 | 12
participants
  Was dose 1 taken? | 15 | 17 | 15 | 16 | 12
  Was dose 2 taken? | 14 | 17 | 3 | 15 | 0

6. Secondary Outcome: Number of Participants in Each Category of the "Subject's Tolerability and Satisfaction Questionaire"
Description: Subject's Tolerability and Satisfaction Questionnaire consists of three questions. Question (Q)1 was "How easy was it to drink the bowel cleanout medicine?" and Q2 was "How did the bowel cleanout medicine taste?". Q3 had five subparts namely: 1. "How often did your tummy hurt since you started the medicine?" and 2. "How often did you feel fullness in your tummy, since you started the cleanout?" and 3. "How often did you wake up last night" and 4. "How often did you feel sick to your stomach (nausea) since you started the cleanout?' and 5. "How much were you bothered by going to the washroom since you started the cleanout?"
  Satisfactory was defined as a response of 1 (Very Easy) or 2 (Easy) on Q1 and a response of 1 (Very Well) or 2 (Well) on Q2.
  Tolerable was defined as a response of 1 (Never) or 2 (Rarely) to the five subparts specified in Q3.
Time Frame: 1 day of colonoscopy
Population: The secondary efficacy analysis was based on the ITT analysis set, which included all participants who were randomized.
Measure: Number; unit: participants
Arm/Group | Prepopik® ½ Sachet x 2 (9-12 Years) | Prepopik® 1 Sachet x 2 (9-12 Years) | Oral Polyethylene Glycol (PEG) Based Preparation (9-12 Years) | Prepopik® 1 Sachet x 2 (13-16 Years) | Oral Polyethylene Glycol (PEG) Based Preparation (13-16 Years)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 14
participants
  Q1-Satisfactory | 9 | 6 | 2 | 8 | 4
  Q2-Satisfactory | 4 | 1 | 5 | 3 | 2
  Q3-Subpart 1-Tolerable | 4 | 9 | 2 | 4 | 5
  Q3-Subpart 2-Tolerable | 9 | 8 | 8 | 7 | 4
  Q3-Subpart 3-Tolerable | 10 | 12 | 11 | 7 | 8
  Q3-Subpart 4-Tolerable | 7 | 9 | 7 | 8 | 3
  Q3-Subpart 5-Tolerable | 9 | 7 | 2 | 5 | 2

ADVERSE EVENTS:
Time Frame: AEs were reported and recorded at Visits 2 (day of randomization) through 5 (Day 28 after the colonoscopy procedure).
Description: Treatment-emergent AE defined as any AE that began during the treatment period (i.e., period during which a participant received an investigational medicinal product) or there was a worsening of a pre-existing medical condition are presented. The results are presented for the safety analysis set.
  One of the participant randomized to Prepopik® ½ sachet x 2 (9-12 years) received Prepopik® 1 sachet x 2 (9-12 years) instead (n=17).
Arm/Group | Prepopik® ½ Sachet x 2 (9-12 Years) | Prepopik® 1 Sachet x 2 (9-12 Years) | Oral Polyethylene Glycol (PEG) Based Preparation (9-12 Years) | Prepopik® 1 Sachet x 2 (13-16 Years) | Oral Polyethylene Glycol (PEG) Based Preparation (13-16 Years)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/17 | 0/15 | 0/16 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17 | 0/15 | 0/16 | 0/12
Other Adverse Events (participants affected / at risk) | 8/15 | 5/17 | 6/15 | 10/16 | 11/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prepopik® ½ Sachet x 2 (9-12 Years) (N=15) | Prepopik® 1 Sachet x 2 (9-12 Years) (N=17) | Oral Polyethylene Glycol (PEG) Based Preparation (9-12 Years) (N=15) | Prepopik® 1 Sachet x 2 (13-16 Years) (N=16) | Oral Polyethylene Glycol (PEG) Based Preparation (13-16 Years) (N=12)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival hemmorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis microscopic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilic colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis eosinophilic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal mucosa hyperemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestinal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot and mouth disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Esophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematocrit decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (2):
  • Study Protocol (2014-07-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT01928862/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT01928862/SAP_001.pdf